CLINICAL TRIAL: NCT01838577
Title: Genetics of EGFR Mutation Study (GEM): a Translational Study of the EORTC Lung Group.
Brief Title: Genetics of EGFR (Epidermal Growth Factor Receptor) Mutation Study
Acronym: GEM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-08114
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: EGFR Mutation Positive Non Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case cohort: Patients with proven EGFR mutation in exons 18-21 from tumor material. Patients with unknown or failed tumor EGFR genotyping will be ineligible. Patients subsequently undergoing re-genotyping which demonstrates an EGFR mutation will become eligible for the "case" cohort.
  No known somatic KRAS, HER2, LKB1, BRAF, or PI3K, mutation or ALK gene rearrangement (or ALK3+ immunohistochemistry). If these mutations are known to be present the patient will be ineligible. However, patients will not be tested specifically for these mutations for this study and patients with unknown status are acceptable. If patients are subsequently tested after enrollment and found to harbor any of these mutations they will be considered ineligible and will be replaced.
  No known Li Fraumeni, Li Fraumeni-like, or Peutz Jeghers syndrome family, or known germline carriers of mutant LKB1 or TP53. Patients will not have to be tested specifically for these syndromes to be eligible for this study.
- Control cohort: Patients known to be somatic EGFR "wild-type," i.e. no mutation detected in exons 18-21 from tumor material.
  Patients with unknown or failed EGFR genotyping will be ineligible. Patients subsequently undergoing re-genotyping which demonstrates an EGFR wild-type will become eligible for the "control" cohort.
  Never smoker (<100 cigarettes in lifetime) or ex-light smoker (stopped ≥1 year ago and smoked ≤10 pack-years).

SUMMARY:
The investigators wish to document the distribution of EGFR somatic mutations, and assess the relationship between specific genotype, clinical demographic, therapy, and survival, in a large cohort of EGFR mutant NSCLC.

The investigators also wish to comprehensively investigate the relationship between germline DNA and risk of EGFR mutant NSCLC developing, through a GWAS (Genome-Wide Association Studies) and candidate gene approach, and explore the relationship between germline DNA and clinical outcome, in order to potentially identify germline genetic modifiers of EGFR TKI (Tyrosine Kinase Inhibitor) outcome.

DETAILED DESCRIPTION:
Objective 1: To identify germline allelic DNA variation associated with somatic EGFR mutation in NSCLC, Objective 2: Correlation between germline allelic variants and survival in EGFR somatic mutant NSCLC.

Objective 3: Study germline allelic DNA variation associated with never /ex light smoking NSCLC.

Objective 4: Catalogue distribution of somatic EGFR mutant genotypes in 1,000 EGFR mutant NSCLC cases and describe their relationship to clinical outcome.

ELIGIBILITY:
* Histologically or cytologically diagnosed NSCLC, all histologies are acceptable.
* Patients can be included in the study with any disease stage and at any time during the disease course.
* Any type (surgery, RadioTherapy, chemotherapy, targeted agents) of previous treatment and any line of treatment are eligible.
* Age ≥18 years.

Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol; those conditions should be discussed with the patient before registration in the trial.

Before patient registration, written informed consent must be given according to ICH/GCP (International Conference on Harmonisation/Good Clinical Practice), and national/local regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case cohort: Patients with proven EGFR mutation in exons 18-21 from tumor material.
  Control cohort: Patients known to be somatic EGFR "wild-type," i.e. no mutation detected in exons 18-21 from tumor material.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-09; Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
For the second objective, the primary endpoint is Overall survival (OS) | 5 years from FPI

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Popat, MD, Principal Investigator — Royal Marsden Hospital, Chelsea, London, UK
Locations (1):
- Royal Marsden, Sutton, United Kingdom